CLINICAL TRIAL: NCT01497535
Title: A Single-centre, Parallel-group, Randomised, Double Blind Trial in Healthy Japanese Subjects Comparing the Within-subject Variability of Insulin Detemir and Insulin Glargine With Respect to Pharmacodynamic and Pharmacokinetic Properties
Brief Title: Within-subject Variability of Insulin Detemir in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN304-1438
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Detemir; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin detemir (Experimental)
  Interventions: Drug: insulin detemir
- Insulin glargine (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin detemir — On four different dosing days where subjects enter a 24-hour euglycaemic glucose clamp procedure, the subject will be allocated to one single dose of either 0.4 U/kg insulin detemir or 0.4 U/kg insulin glargine administered subcutaneously (s.c., under the skin)
  Arms: Insulin detemir
Drug: insulin glargine — On four different dosing days where subjects enter a 24-hour euglycaemic glucose clamp procedure, the subject will be allocated to one single dose of either 0.4 U/kg insulin detemir or 0.4 U/kg insulin glargine administered subcutaneously (s.c., under the skin)
  Arms: Insulin glargine

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare the within-subject variability of insulin detemir to that of another basal insulin analogue, insulin glargine in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese men or women
* Holding a Japanese pass-port and Japanese-born parents
* Considered generally healthy upon completion of medical history and physical examination as judged by the Investigator
* Body Mass Index (BMI) between 18 and 30 kg/m^2, incl.
* Fasting blood glucose maximum 6 mmol/L

Exclusion Criteria:

* Clinically significant abnormal haematology or biochemistry screening tests, as judged by the Investigator
* Any serious systemic infectious disease that occurred during the four weeks prior to the first dose of the trial product, as judged by the Investigator
* Subject with history of alcohol or drug dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-05-27 (Actual); Primary Completion 2004-10-31 (Actual); Study Completion 2004-10-31 (Actual)

PRIMARY OUTCOMES:
Maximum glucose infusion rate (GIRmax)

SECONDARY OUTCOMES:
Area under the glucose infusion rate curve (AUCGIR)
Time to maximum glucose infusion rate (tGIRmax)
Area under the insulin concentration curve (AUC)
Maximum insulin concentration (Cmax)
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com